CLINICAL TRIAL: NCT04020887
Title: A Proof-of-concept Observational Study Evaluating the Acceptability and Utility of a Telemedicine Solution for the Post Anesthesia Care Unit
Brief Title: Telemedicine Control Tower for the Post-Anesthesia Care Unit
Acronym: PACU Telemed
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Michael Avidan, Professor of Anesthesiology and Surgery, Washington University School of Medicine
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 201901180
Record Dates: First submitted 2019-03-06; First posted 2019-07-16 (Actual); Results first posted 2023-07-19 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2021-12

CONDITIONS: Elective Surgery
Keywords: Telemedicine; Post Anesthesia Care Unit (PACU)

STUDY DESIGN:
Intervention Model Description: The first phase is an observation phase and the next phase is an interaction phase.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Observation Phase (No Intervention): In the first three months of this proof-of-concept study, a telemedicine center for the PACU will monitor patients assigned to PACU bays. Both telemedicine center clinicians and nurses caring for patients in these PACU bays will independently record information on patient physiological derangements, treatable symptoms, situations requiring urgent medical intervention, and discharge readiness (based on the modified Aldrete scale). During this phase of the study, clinicians in the telemedicine center will not communicate with clinicians in the PACU (nurses or physicians), unless there was a patient safety event.
- Interaction Phase (Experimental): In the three months following the observation phase, clinicians in the telemedicine center will interact with clinicians and patients in the two designated PACU bays using audio-visual technology. The clinicians in the telemedicine center will continue to document information on physiological derangements, treatable symptoms, situations requiring urgent medical intervention, and discharge readiness.
  Interventions: Device: Alertwatch - Interaction

INTERVENTIONS:
Device: Alertwatch - Interaction — Decision-support software, customized for the PACU environment, Interaction between the telemedicine center and the PACU
  Arms: Interaction Phase

SUMMARY:
A single center prospective before-and-after proof-of-concept study to evaluate a telemedicine center for the PACU.

DETAILED DESCRIPTION:
A proof-of-concept study in perioperative telemedicine that aims to demonstrate the (i) acceptability and (ii) utility of integrating telemedicine into the PACU environment. This proof-of-concept study will be conducted in the PACU.

ELIGIBILITY:
Adults (age ≥ 18) undergoing elective surgery at Barnes Jewish Hospital in St. Louis, Missouri will be enrolled

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-12-06 (Actual); Study Completion 2021-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Avidan, MBBcH, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Derived] Budelier TP, King CR, Goswami S, Bansal A, Gregory SH, Wildes TS, Abraham J, McKinnon SL, Cooper A, Kangrga I, Martin JL Jr, Milbrandt M, Evers AS, Avidan MS. Protocol for a proof-of-concept observational study evaluating the potential utility and acceptability of a telemedicine solution for the post-anesthesia care unit. F1000Res. 2020 Oct 20;9:1261. doi: 10.12688/f1000research.26794.1. eCollection 2020. PMID 33214879

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Observation Phase | Interaction Phase
Started | 304 | 256
Completed | 304 | 256
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Observation Phase | Interaction Phase | Total
Number analyzed (Participants) | 304 | 256 | 560
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.9 (15.7) | 55.7 (15) | 55.8 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 194 | 157 | 351
  Male | 110 | 99 | 209
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 6 | 11
  Not Hispanic or Latino | 295 | 248 | 543
  Unknown or Not Reported | 4 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 0 | 3
  Asian | 4 | 4 | 8
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 64 | 49 | 113
  White | 230 | 201 | 431
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 304 | 256 | 560
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 30.7 (8.6) | 31.5 (9.9) | 31.0 (9.2)
ASA Physical Status [Count of Participants; unit: Participants] — Range, 1 to 6; 1 indicates healthy, 2 indicates mild systemic disease, 3 indicates severe systemic disease, 4 indicates severe systemic disease that is a constant threat to life, 5 indicates not expected to survive without surgery, 6 indicates neurologically deceased organ donor. In this study, only patients with an ASA 1 to 5 were collected.
  Participants
    ASA 1 | 10 | 9 | 19
    ASA 2 | 157 | 127 | 284
    ASA 3 | 129 | 119 | 248
    ASA 4 | 8 | 1 | 9
    ASA 5 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Difference in Time to PACU Discharge Determination From Observation to Interaction Phase
Description: The difference in discharge readiness time between the observation and interaction phases will be compared
Time Frame: up to 1 day
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | Observation Phase | Interaction Phase
Number analyzed (Participants) | 304 | 256
Minutes | 84.5 [54.0 to 116.5] | 91.5 [62.0 to 145.0]
Statistical Analysis 1: Comparison: Observation Phase vs Interaction Phase; Difference in time to PACU discharge determination from observation to interaction phase [ Time Frame: 6 months]: The difference in discharge readiness time between the observation and interaction phases will be compared; Test type: Superiority; Median Difference (Final Values) = 6.0, 95% CI 2-sided [-6.01 to 18.01]

2. Secondary Outcome: Demonstrate the Potential Ability of a Remote Telemedicine Center for the PACU to Assist With PACU Functions.
Description: Percent of patients the telemedicine center participated in the hand-off process from OR to the PACU in both the observation and interaction phases. Participation by the telemedicine center was successful if the telemedicine center could both remotely join the hand-off process and collect relevant patient care information.
Time Frame: up to 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Observation Phase | Interaction Phase
Number analyzed (Participants) | 304 | 256
Participants
  Hand-off participation Yes | 205 | 249
  Hand-off participation No | 99 | 7
Statistical Analysis 1: Comparison: Observation Phase vs Interaction Phase; Test type: Superiority; Difference Between Proportions = 29.80, 95% CI 2-sided [23.82 to 35.66]

3. Secondary Outcome: Detection of Physiological Derangements in PACU Patients
Description: The proportion of physiological derangements identified in the telemedicine center in both the observation and interaction phases
Time Frame: approximately 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Observation Phase | Interaction Phase
Number analyzed (Participants) | 304 | 256
Participants | 39 | 26
Statistical Analysis 1: Comparison: Observation Phase vs Interaction Phase; Test type: Superiority; Difference Between Proportions = -2.67, 95% CI 2-sided [-8.18 to 3.02]

4. Secondary Outcome: Identification of Symptoms Requiring Treatment in PACU Patients
Description: Number of patients identified with symptoms requiring treatment in PACU such as pain or nausea in both the observation and interaction phases
Time Frame: approximately 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Observation Phase | Interaction Phase
Number analyzed (Participants) | 304 | 256
Participants | 72 | 94
Statistical Analysis 1: Comparison: Observation Phase; Test type: Superiority; Difference Between Proportions = 13.03, 95% CI 2-sided [5.16 to 20.79]

5. Secondary Outcome: Recognition of Situations Requiring Emergency Medical Intervention
Description: The number of patients identified requiring emergency medical intervention in both the observation and interaction phases
Time Frame: approximately 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Observation Phase | Interaction Phase
Number analyzed (Participants) | 304 | 256
Participants | 2 | 3
Statistical Analysis 1: Comparison: Observation Phase vs Interaction Phase; Test type: Superiority; Difference Between Proportions = 0.51, 95% CI 2-sided [-1.63 to 3.07]

6. Secondary Outcome: Determination of Patient Readiness for PACU Discharge
Description: Number of patients determined to be ready for PACU discharge prior to documentation by the PACU Team in both the observation and interaction phases
Time Frame: approximately 1 day
Population: For cases where patients were discharged from the PACU during ePACU operational hours (M-F; 0700- 1600).
Measure: Count of Participants; unit: Participants
Arm/Group | Observation Phase | Interaction Phase
Number analyzed (Participants) | 260 | 204
Participants | 233 | 199
Statistical Analysis 1: Comparison: Observation Phase vs Interaction Phase; Test type: Superiority; Difference Between Proportions = 7.9, 95% CI 2-sided [3.13 to 12.71]

ADVERSE EVENTS:
Time Frame: approximately 1 day
Arm/Group | Observation Phase | Interaction Phase
All-Cause Mortality (participants affected / at risk) | 0/304 | 0/256
Serious Adverse Events (participants affected / at risk) | 0/304 | 0/256
Other Adverse Events (participants affected / at risk) | 0/304 | 0/256

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-26): https://cdn.clinicaltrials.gov/large-docs/87/NCT04020887/Prot_SAP_000.pdf